CLINICAL TRIAL: NCT07200128
Title: Satisfaction and Treatment Experiences With RitlEcitiNib And Traditional Treatments for Severe Alopecia Areata Among Adults in the United States (SERENATA)
Brief Title: A Study to Learn About the Medicine Called Ritlecitinib in Adults With Severe Alopecia Areata in Real-world Settings
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7981115
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Severe Alopecia Areata
Keywords: Ritlecitinib; Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with severe Alopecia Areata
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — As provided in real world practice

SUMMARY:
This study is a secondary analysis of the Adelphi Real World Alopecia Areata II United States Disease Specific Programmes database. This database contains data from a cross-sectional study capturing linked physician and patient survey data for dermatologists who treat alopecia areata and patients diagnosed with alopecia areata in the United States. The retrospective analysis of these data will evaluate experiences of patients and dermatologists receiving/prescribing ritlecitinib for severe alopecia areata in the United States. Specifically, the study will describe characteristics of patients who received ritlecitinib for severe alopecia areata, including demographics, clinical characteristics at the time of starting ritlecitinib, and their alopecia areata-related treatment history. The study will also report dermatologist satisfaction with treatment and change in the patient's alopecia areata severity and disease activity from the start of ritlecitinib to different time points on treatment.

ELIGIBILITY:
Aged 18 years or older with severe alopecia areata

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe AA treated with ritlecitinib by dermatologists in the US.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
% of patients for whom their clinician was "satisfied" with current control of alopecia areata | 11/15/2023 to 06/10/2024
% of patients with clinician-assessed mild, moderate, or severe disease | 11/15/2023 to 06/10/2024
% of patients with clinician assessed progressive, stable, or improving disease | 11/15/2023 to 06/10/2024

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981115